CLINICAL TRIAL: NCT05869890
Title: Ureteroscopic Laser Modality on Total Lasing Time and Total Energy in Patients With Large, Dense Renal Calculi
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the institution
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Brenda Romeo, Research Manager for Luay Alshara, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6286
Record Dates: First submitted 2023-05-12; First posted 2023-05-22 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Renal Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Flexible Ureteroscopy with Dusting (Other): Flexible ureteroscopy with the dusting lasing technique. MOSES parameters will be set to an energy of 0.3-0.4 Jules and a frequency of 50-80 hertz
  Interventions: Device: MOSES laser system
- Flexible Ureteroscopy with Fragmentation (Other): Flexible ureteroscopy utilizing the Fragmentation lasing technique. MOSES parameters will be set to 0.8-1 JULES and a frequency of 8-10 hertz
  Interventions: Device: MOSES laser system
- Flexible Ureteroscopy with Hybrid (Other): Flexible ureteroscopy utilizing the Hybrid lasing technique which will use both sets of parameters.
  Interventions: Device: MOSES laser system

INTERVENTIONS:
Device: MOSES laser system — A holmium laser technology widely used as the gold standard for laser lithotripsy for ureteroscopy treatment of renal calculi,

SUMMARY:
This study will examine the effects of ureteroscopic lasing technique (dusting, fragmentation and a hybrid approach) on total lasing time and total energy in patients with a large renal calculi burden of single or multiple stones with the sum of its longest diameters between 10-20 mm and having mean Hounsfield units of 1000 or more.

DETAILED DESCRIPTION:
This study will examine the effects of ureteroscopic lasing technique (dusting, fragmentation and a hybrid approach) on total lasing time and total energy in patients with a large renal calculi burden of single or multiple stones with the sum of its longest diameters between 10-20 mm and having mean Hounsfield units of 1000 or more. Additionally, we will observe the impact of these parameters on total operative time.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-80.
* Any gender, race or ethnicity may be included- these factors play a small, if any role on renal calculi formation and ability to withstand procedure.
* Must be suitable for a flexible ureteroscopy as determined by the MD
* Large renal calculi burden of single or multiple stones with the sum of its longest diameters between 10-20 mm
* An average stone density of at least 1000 Hounsfield units.

Exclusion Criteria:

* Those with a stone burden less than 10mm or more than 20mm.
* Those with an average stone density below 1000 Hounsfield units.
* Patients who are dependent on mandatory anticoagulation therapies and cannot stop for surgery
* Patients that cannot undergo ureteral access sheath placement
* Patients with abnormal anatomy such as horseshoe kidney
* Patients with a history of:

  * Ipsilateral upper urinary tract reconstructive procedures on the side of the renal calculi
  * Ipsilateral ureteral strictures
  * Prior radiotherapy of the abdomen or pelvis
  * Neurogenic bladder
  * Spinal cord injuries
  * Those who are pregnant
  * Currently being treated for infection or cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Reduced OR time | 2 hours
  Hybrid technique will result in overall reduced OR time
Less Energy Transmission to Patient | 2 hours
  Hybrid technique will have less energy transmission to the patient

SECONDARY OUTCOMES:
Stone Free | 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical College, Albany, New York, United States